CLINICAL TRIAL: NCT03472755
Title: Subjective Walking Capacity : Comparison of Direct Anterior and Posterior Surgical Approaches in Regards to the Patient' Physical Characteristics (MOPHEM)
Brief Title: Comparison of Direct Anterior and Posterior Surgical Approaches in Regards to the Patient' Physical Characteristics
Acronym: MOPHEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in setting up the study in the investigator site
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2017_843_0023
Record Dates: First submitted 2018-02-05; First posted 2018-03-21 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Hip Arthropathy
Keywords: hip arthroplasty; surgeries; physical fitness; perception; energetic cost; autonomy

STUDY DESIGN:
Intervention Model Description: Patients provided written informed consent to participate in this study, as approved by the local ethics committee. Prior to surgery, patients were informed about the benefits and risk of the conventional posterolateral and direct anterior approaches. Then they performed postural test and a Performance-Oriented Mobility Assessment Walking test with and without step. After randomization, patients were operated according the conventional posterolateral or direct anterior techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The posterolateral approach (Other): The posterolateral approach was used for implantation among patients in lateral position. This approach goes through the gluteus maximus, the piriformis and superior gemeli muscles are detached and later reattached to bone
  Interventions: Other: The posterolateral approach
- Direct anterior techniques. (Other): . In the direct anterior technique, patients were fixed in a supine position, a small entry incision was made in the vessel free interval between the tensor fasciae latae and the sartorius muscles and the prosthesis socket were put in place. Via a second dorsal incision, after releasing the external rotators, the prosthesis stem and ball were implanted and the two parts of the prosthesis were attached.
  Interventions: Other: Direct anterior technique

INTERVENTIONS:
Other: The posterolateral approach — The posterolateral approach was used for implantation among patients in lateral position. This approach goes through the gluteus maximus, the piriformis and superior gemeli muscles are detached and later reattached to bone
  Arms: The posterolateral approach
Other: Direct anterior technique — patients were fixed in a supine position, a small entry incision was made in the vessel free interval between the tensor fasciae latae and the sartorius muscles and the prosthesis socket were put in place. Via a second dorsal incision, after releasing the external rotators, the prosthesis stem and ball were implanted and the two parts of the prosthesis were attached
  Arms: Direct anterior techniques.

SUMMARY:
Recent increased interest in tissue-sparing and minimally invasive arthroplasty has given rise to a sharp increase in the utilization of direct anterior total hip arthroplasty.

DETAILED DESCRIPTION:
* Purpose: The direct anterior approach to the hip has been suggested to have several advantages compared to previously classical approaches. However, no studies focused on the effects of these different surgeries on patients' perception recovery and walking efficiency according the initial physical fitness. Therefore, the purpose of this study is to compare the effects of surgical procedures on perceptual walking skills and efficiency according to the patients' physical fitness.
* Abstract : Some earlier studies report differences between surgery types in self- reported mobility, functional recovery and residual hip pain. The direct anterior approach to the hip has been suggested to have several advantages compared to previously popular approaches through its use of an intra-muscular and intra-nervous interval between the tensor fasciae latae and sartorius muscles. However, patients' physical fitness, postural response and perceptual walking skill relation was not taking account. 80 patients will be tested, one before and at various times after hip surgery. In randomized conditions, our patients will be divided in two groups, according the surgery approaches and their physical fitness. All patients performed a Performance-Oriented Mobility Assessment Walking test with and without step and the PMA, Harris, Oxford 12 and Womac scores will be evaluated before, 3 weeks, 6 weeks, 3 months and 1 year after the surgery. During the Performance-Oriented Mobility Assessment Walking test, self-reported walking capacity, rating of exertion perception and walking parameters will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Body mass index < 35
* Scheduled hip arthroplasty surgery
* Exclusion Criteria:
* No health coverage
* Age > 85 years
* Body mass index ≥ 35
* Cognitive impairment (score Mini Mental Statue < 24)
* Any other osteo-articular diseases than the operated hip, any muscular or neurological diseases that could penalize the walk

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-23 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01-20 (Estimated)

PRIMARY OUTCOMES:
hip's range of motion. | 1 year